CLINICAL TRIAL: NCT01284192
Title: A Phase 1, Multicenter, Open-Label, Dose Escalation Study of ASP3026 in Subjects With Advanced Malignancies
Brief Title: Study of an Investigational Drug, ASP3026, in Patients With Advanced Malignancies (Solid Tumors and B-Cell Lymphoma)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A3026-CL-0101
Record Dates: First submitted 2011-01-25; First posted 2011-01-26 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Advanced Malignancies; Positive for Anaplastic Lymphoma Kinase; Positive for Proto-Oncogene Tyrosine-Protein Kinase ROS; Solid Tumor; B-Cell Lymphoma
Keywords: B-cell Lymphoma; Advanced Malignancies; Anaplastic Lymphoma Kinase (ALK); ASP3026; Solid Tumor
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — ASP3026

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ASP3026 (Experimental): Subjects will receive escalated doses of ASP3026 to determine the maximum tolerated dose (MTD)
  Interventions: Drug: ASP3026

INTERVENTIONS:
Drug: ASP3026 — Tablet

SUMMARY:
This study is to evaluate the safety and anti-tumor activity of ASP3026 in patients with advanced malignancies (solid tumors and B-cell lymphoma).

DETAILED DESCRIPTION:
This study will be conducted using a traditional 3 + 3 dose escalation study design. Enrollment of at least 3 subjects is planned for each dosing cohort until the Maximum Tolerated Dose (MTD) is determined. Up to three additional subjects per cohort may be enrolled if each additional subject is known to be positive for Anaplastic Lymphoma Kinase (ALK) or Proto-Oncogene Tyrosine-Protein Kinase ROS (ROS) abnormalities. The decision to expand a cohort or dose escalate will be based on the occurrence of dose limiting toxicities (DLTs) in Cycle 1 that are considered by the Investigator to be related (possibly or probably) to ASP3026. Intra-subject dose escalation will be allowed at the discretion of the investigators. The Safety Data Review Committee may elect to enroll additional subjects in a cohort to further evaluate the dose level. Once the MTD is determined, approximately 20 additional subjects with Anaplastic Lymphoma Kinase (ALK) abnormalities will be enrolled at the Recommended Phase 2 Dose. Each cycle will include 28 days of continuous dosing with ASP3026. Treatment with ASP3026 may continue until one of the discontinuation criteria is met.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Histologically or cytologically confirmed diagnosis of a relapsed/refractory solid tumor or B-cell lymphoma and meets at least 1 of the following criteria:

  * Disease progression despite standard therapies
  * No standard therapies are available or such therapies are not anticipated to result in a durable response
  * Standard therapies are considered unsuitable or have been refused
* Able to take oral medications
* Life expectancy > 12 weeks
* For the expansion cohort of the study, all subjects must be confirmed to be positive for ALK gene abnormalities
* Subjects with stable brain metastasis will be allowed

Exclusion Criteria:

* Active central nervous system (CNS) metastases or leptomeningeal involvement as assessed through medical history review and physical examination (dose escalation subjects only)
* Known history of a positive test for hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV)
* Known hereditary or acquired immunodeficiency syndrome or human immunodeficiency virus (HIV) infection
* Cardiac arrhythmias > Grade 1 using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v. 4.03
* Class 3 or 4 New York Heart Association congestive heart failure, acute coronary syndrome, myocardial infarction or cerebrovascular accident within 6 months prior to Cycle 1, Day 1
* Inadequate bone marrow, renal, and/or hepatic function
* Confirmed active peptic ulcer disease or history of gastrointestinal bleeding within the past 3 months
* Known history of long QT syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-12; Primary Completion 2014-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ASP3026 assessed by recording of adverse events, laboratory assessments, vital signs, electrocardiograms (ECGs) and clinical observations | Up to 30 days after last subject discontinues treatment

SECONDARY OUTCOMES:
Pharmacokinetic assessment through analysis of blood and urine samples | Up to Day 29
Objective response rate (ORR) | 30 Days after the last subject discontinues treatment
  Objective response rate is the proportion of subjects who experience complete response/remission (CR) or partial response/remission (PR)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development
Locations (6):
- United States (6):
  - Site US160, Orange, California
  - Site US184, Sacramento, California
  - Site US11, Chicago, Illinois
  - Site US2688, Detroit, Michigan
  - Site US2492, Houston, Texas
  - Site US1905, San Antonio, Texas

REFERENCES:
- [Derived] Li T, LoRusso P, Maitland ML, Ou SH, Bahceci E, Ball HA, Park JW, Yuen G, Tolcher A. First-in-human, open-label dose-escalation and dose-expansion study of the safety, pharmacokinetics, and antitumor effects of an oral ALK inhibitor ASP3026 in patients with advanced solid tumors. J Hematol Oncol. 2016 Mar 10;9:23. doi: 10.1186/s13045-016-0254-5. PMID 26966027